CLINICAL TRIAL: NCT02387658
Title: Outcomes in Femoropopliteal Disease Stratified by Translesional Pressure Gradient
Status: Completed | Type: Observational
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Subhash Banerjee, Chair of Cardiology North Texas VA Medical Center, North Texas Veterans Healthcare System
Other Study IDs: Dallas VA IRB Protocol #14-076
Record Dates: First submitted 2015-03-08; First posted 2015-03-13 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Peripheral Arterial Disease; Claudication
Keywords: peripheral arterial disease; claudication; translesional pressure gradient; pressure wire; six minute walk; superficial femoral artery; pressure gradient; endovascular
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- final TLG </=11 mmHg: includes all patients who have a final mean translesional gradient measurement (TLG) < 11 mmHg regardless if revascularization is done or not.
  Interventions: Procedure: translesional gradient measurement
- final TLG > 11 mmHg: includes all patients who have a final mean translesional gradient measurement (TLG) > 11 mmHg regardless if revascularization is done or not.
  Interventions: Procedure: translesional gradient measurement

INTERVENTIONS:
Procedure: translesional gradient measurement — Patients will be stratified into two groups based on the final mean translesional pressure gradient obtained in the femoropopliteal arterial bed after revascularization or just after angiography if no revascularization is done.

SUMMARY:
1. To perform an observational analysis to determine if mean translesional gradient measurements (TLG) are associated with differences in clinical outcomes in patients with femoropopliteal arterial disease and claudication.
2. Hypothesis: Patients stratified by a residual translesional gradient </= 11 mmHg after peripheral revascularization or angiography alone will have better clinical outcomes than patients with TLG > 11 mmHg as assessed by six minute walk (6MW), walking impairment questionnaire scores (WIQ), ankle brachial index and need for repeat procedure at 6 months.

DETAILED DESCRIPTION:
The role of measuring translesional pressure gradients(TLG) in peripheral arterial disease lesions below the iliac artery is unclear. In a previous study the investigators demonstrated that a pressure wire can be effectively used to measure gradients in the femoropopliteal (FP) arterial bed showing good correlation between TLGs recorded with exercise ankle brachial index and walking impairment scores. However there is a no evidence that effectively modifying the gradient or having a high residual gradient after revascularization or just with medical therapy correlates with worse clinical outcomes.

This is a prospective, single center, observational clinical study to evaluate whether measurement of mean residual TLG at the time of angiography and/or immediately after endovascular revascularization are associated with clinically important outcomes in patients with claudication symptoms.

Prior to angiography they will be asked to complete an ankle brachial index evaluation, baseline six minute walk test and walking impairment questionnaire. Arterial access should be obtained in the contralateral common femoral artery to the symptomatic limb if feasible. Angiographic images are to be obtained, interpreted and clinical decisions regarding endovascular treatment are to be made per treating physician's discretion prior to obtaining translesional pressure gradients. In patients whose angiogram does not meet exclusion criteria and do not have a chronic total occlusion (CTO) a baseline TLG will be obtained. A 0.014" pressure wire/catheter to measure pressure will be inserted. After baseline calibration in the superficial femoral artery, the wire will be inserted past the narrowest lesion into the popliteal vessel. Intra-arterial adenosine 100-200 mcg will be given for hyperemia and measurements are to be recorded. If an intervention is planned, repeat measurements are to be obtained at the end of the procedure. If no intervention is planned this will be the residual or final TLG recorded. If baseline measurement are unable to obtained due to a CTO then only a post intervention residual TLG will be obtained and included in analysis. The operator will be blinded to the pre and post TLG measurements by turning the display monitor away from the procedure table and towards the recorder situated in the procedure room when measurements are being obtained.

Patients will follow up within two weeks post angiography for routine scheduled follow up and will obtain repeat ABI, WIQ, and six minute walk if they underwent revascularization. Treating physicians and study coordinators collecting these test measurements will be blinded to TLG measurements but not to angiography and treatment. Patients will again be evaluated at 6 months follow up with repeat ABI, WIQ and six minute walk.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* At least 18 years old
* Unilateral lower limb claudication Rutherford class 2-4
* Subjects must be able to complete screening six minute walk, walking impairment questionnaire, and baseline ankle brachial index
* Estimated survival ≥1 year in the judgment of the primary operator
* Documented symptomatic femoropopliteal (FP) atherosclerotic disease with at least moderate angiographic stenosis in the symptomatic lower extremity
* Subjects with multilevel disease can be screened and enrolled after treatment of other non FP PAD

Exclusion Criteria:

* Life expectancy less than 12 months or other medical co-morbid condition(s) that could limit the subject's ability to participate in the trial, limit the subject's compliance with the follow-up requirements, or impact the scientific integrity of the trial
* Severe Bilateral claudication
* Known hypersensitivity or contraindication to contrast dye that, in the opinion of the investigator, cannot be adequately pre-medicated
* Known hypersensitivity to adenosine or moderate to severe asthma
* Pregnancy
* Serum Creatinine >2.5
* Vascular graft, aneurysm or postsurgical stenosis of the target vessel
* Documented untreated severe iliac or below-the knee stenosis with < 2 vessel run-off in leg with femoropopliteal stenosis or untreated bilateral symptomatic peripheral arterial disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with claudication symptoms and femoropopliteal disease referred for peripheral angiography and possible revascularization.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-02-06 (Actual); Primary Completion 2016-07-13 (Actual); Study Completion 2016-07-13 (Actual)

PRIMARY OUTCOMES:
Change in six minute walk distance in meters at 6 months | 6 months +/- 15 days after enrollment
  Compare change in six minute walk distance at 2 weeks post angiography +/- revascularization to distance walked at 6 months +/- 15 days between patients stratified by a residual mean translesional gradient > 11 mmHg or </= 11 mmHg. The six minute walk test involves walking in a straight 100m hallway back and forth for as far as possible during a six minute time span.

SECONDARY OUTCOMES:
Change Walking Impairment Questionairre (WIQ)Score at 6 months | 6 months +/- 15 days after enrollment
  Compare change in WIQ scores from within 2 weeks post angiography +/- revascularization to WIQ score at 6 months +/- 15 days between patients stratified by a residual mean translesional gradient > 11 mmHg or </= 11 mmHg . The walking impairment score used is based on the patient completing short questionnaire about perceived degree of walking impairment at various distances.
Change in Ankle Brachial Index (ABI) at 6 months | 6months +/- 15 days after enrollment
  Change in ABI between patients stratified by a residual mean translesional gradient > 11 mmHg or </= 11 mmHg from the index within 2 weeks post TLG measurement to index at 6 months after measurement
Change in six minute walk distance from baseline to within 2 weeks post revascularization | baseline pre revascularization to two weeks post measurement
  Change in six minute walk from baseline measurement in those patients that undergo revascularization to six minute walk distance checked within 2 weeks after revascularization.
Change in WIQ score from baseline to within 2 weeks post revascularization | baseline pre revascularization to two weeks post measurement
  Change in WIQ score from baseline measurement in those patients that undergo revascularization to six minute walk distance checked within 2 weeks after revascularization.
Need for repeat revascularization or amputation as assessed by rates of need in repeat revascularization or amputation | six months
  compare rates of need in repeat revascularization or amputation between patients stratified by a residual mean translesional gradient > 11 mmHg or </= 11 mmHg during 6 month period after TLG measurement.

OTHER OUTCOMES:
Secondary analysis evaluating correlation between change in 6 minute walk distance at 6 month and residual translesional gradients. | 6 months
  evaluate for linear correlation between change in six minute walk from baseline to 6 months to mean translesional gradient
Secondary analysis evaluating correlation in change in WIQ score at 6 month and residual translesional gradients. | 6 months
  evaluate for linear correlation between change in WIQ from baseline to 6 months to mean translesional gradient

CONTACTS AND LOCATIONS:
Locations (1):
- VA North Texas Health Care System, Dallas, Texas, United States

REFERENCES:
- [Background] Klein AJ, Pinto DS, Gray BH, Jaff MR, White CJ, Drachman DE; Peripheral Vascular Disease Committee for the Society for Cardiovascular Angiography and Interventions. SCAI expert consensus statement for femoral-popliteal arterial intervention appropriate use. Catheter Cardiovasc Interv. 2014 Oct 1;84(4):529-38. doi: 10.1002/ccd.25504. Epub 2014 Jun 12. PMID 24753020
- [Background] Walker C. What is the role of translesional pressure gradient measurement in peripheral intervention? J Invasive Cardiol. 2011 Sep;23(9):357. No abstract available. PMID 21891804
- [Background] Archie JP Jr. Analysis and comparison of pressure gradients and ratios for predicting iliac stenosis. Ann Vasc Surg. 1994 May;8(3):271-80. doi: 10.1007/BF02018175. PMID 8043361
- [Background] Banerjee S, Badhey N, Lichtenwalter C, Varghese C, Brilakis ES. Relationship of walking impairment and ankle-brachial index assessments with peripheral arterial translesional pressure gradients. J Invasive Cardiol. 2011 Sep;23(9):352-6. PMID 21891803
- [Background] Garcia LA, Carrozza JP Jr. Physiologic evaluation of translesion pressure gradients in peripheral arteries: comparison of pressure wire and catheter-derived measurements. J Interv Cardiol. 2007 Feb;20(1):63-5. doi: 10.1111/j.1540-8183.2007.00213.x. PMID 17300406
- [Background] De Bruyne B, Manoharan G, Pijls NH, Verhamme K, Madaric J, Bartunek J, Vanderheyden M, Heyndrickx GR. Assessment of renal artery stenosis severity by pressure gradient measurements. J Am Coll Cardiol. 2006 Nov 7;48(9):1851-5. doi: 10.1016/j.jacc.2006.05.074. Epub 2006 Oct 17. PMID 17084261
- [Background] Belch JJ, Topol EJ, Agnelli G, Bertrand M, Califf RM, Clement DL, Creager MA, Easton JD, Gavin JR 3rd, Greenland P, Hankey G, Hanrath P, Hirsch AT, Meyer J, Smith SC, Sullivan F, Weber MA; Prevention of Atherothrombotic Disease Network. Critical issues in peripheral arterial disease detection and management: a call to action. Arch Intern Med. 2003 Apr 28;163(8):884-92. doi: 10.1001/archinte.163.8.884. No abstract available. PMID 12719196
- [Background] Tetteroo E, van Engelen AD, Spithoven JH, Tielbeek AV, van der Graaf Y, Mali WP. Stent placement after iliac angioplasty: comparison of hemodynamic and angiographic criteria. Dutch Iliac Stent Trial Study Group. Radiology. 1996 Oct;201(1):155-9. doi: 10.1148/radiology.201.1.8816537.